CLINICAL TRIAL: NCT05100888
Title: Theta-burst rTMS in Schizophrenia to Ameliorate Negative and Cognitive Symptoms: a Double-blind, Randomized Clinical Trial
Brief Title: Theta-burst rTMS in Schizophrenia to Ameliorate Negative and Cognitive Symptoms
Acronym: tbTMS_SCH21
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Gábor Csukly, Assistant Professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TB-rTMS_SCH2021
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Transcranial Magnetic Stimulation Repetitive; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theta-burst rTMS (Experimental): Theta-burst repetitive transcranial magnetic stimulation
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham stimulation (Sham Comparator): Sham stimulation of the same location
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — Theta-burst stimulation

SUMMARY:
The major target of the study is to confirm the safety and efficacy of our augmented protocol of theta-burst TMS in schizophrenia. Our aim is to confirm the beneficial effects of rTMS treatment on multiple aspects of the disorder such as (1) clinical aspect in terms of PANSS, (2) cognitive aspect such as emotion recognition (ER) and working memory (WM) / distractor filtering (DF) performance, and (3) neurobiology in terms of electrophysiology correlates of ER, WM and DF such as event related theta synchronization, resting state theta power, and network connectivity. Response prediction to (theta-burst) TB-rTMS will be the exploratory part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of schizophrenia or schizoaffective disorder;
2. clinically stabilized on antipsychotic: a stable dose of antipsychotic medication for >4 weeks;
3. age 18-55 years, and
4. presence of negative symptoms (based on PANSS): a negative subscore ≥16 points and [one of items N1-N7 scoring ≥4 or two items N1-N7 scoring ≥3]

Exclusion Criteria:

1. any significant neurological illness;
2. mental retardation
3. history of head injury with loss of consciousness for more than 1 hour
4. history of epileptic seizures or epileptic activity on the baseline EEG (evaluated by an expert in clinical EEG and epilepsy),
5. alcohol or drug abuse within the past 3 months, and
6. depressive episode or antidepressant treatment in the past 4 weeks.
7. Severe positive symptoms inferfere with cognitive tests
8. ECT in the medical history
9. Implanted pacemaker, implanted drug pump, cochlear implant, implanted defibrillator, implanted neurostimulator or any other TMS incompatible implanted metal device
10. Skin surface is severly injured in the stimulated region of the skull
11. Sclerosis multiplex
12. Pregnancy
13. Severe sleep deprivation
14. Severe heart failure
15. Increased intracranial pressure
16. Untreated migrain

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale, Negative subscore | 4 weeks
  The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia. It is the gold standard in the treatment monitoring of schizophrenia.The scale has three subscales : positive, negatve and general symptom score. We use the negative subscore as primary outcome. Its minimum and maximum scores are 7 and 49 respectively. Higher values indicate worse outcome.

SECONDARY OUTCOMES:
Cognitive functioning/Short-Term Memory - The Digit Span Forward and Backward tests | 4 weeks
  They will be used to assess working memory. Digits Recalled is the primary outcome measure ranging between 2 and 10. Lower values indicate worse outcome.
Cognitive functioning/Executive functioning - Wisconsin Card Sorting test | 4 weeks
  The test will be used to measure cognitive flexibility/Executive functioning. Number of persevarative errors is the major outcome variable of the test, its minimum is 0, while it has no theroretical maximum value. Higher values indicate worse outcome. Punishment sensitivity (P) from the reinforcement learning model of WCST will also be used as outcome variable. Its minimum value is 0 and it has no theoretical maximum value. Lower values indicate worse outcome.
Social cognition 1 - The Baron-Cohen 'Reading the Mind in the Eyes Test ' | 4 weeks
  The total score is the primary outcome, which ranges between 0 and 37 points. Lower values indicate worse outcome.
Social cognition 2 - The 'Faux Pas' test. | 4 weeks
  Measures Theory of Mind (ToM), and the primary outcome measure is the total score, which ranges between 0 and 1. Lower values indicate worse outcome.
Facial Emotion Recogniton - Karolinska Directed Emotional Face set | 4 weeks
  Facial expression recognition task. Subject have to identify emotional expressions from photographs of 8 male and 8 female subjects. The pictures are chosen from Karolinska Directed Emotional Face set. There are 3 photographs from each faces (happy, neutral, and sad). Hit rate is the primary outcome measure, which ranges from 0% to 100%, and lower values indicate worse outcome. A 64-channel high-density EEG is recorded during the task, and ERPs (e.g., n170) are calculated for each emotion condition and EEG channel.
Safety in terms of adverse events | 4 weeks
  Safety in terms of the number of serious adverse events (SAE).
  A Serious Adverse Event is any untoward medical occurrence that:
  * Results in death
  * Is life-threatening or
  * Requires in-patient confinement or prolongation of existing confinement or
  * Results in persistent or significant disability/incapacity or
  * Is a congenital anomaly/birth defect.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Budapest, Budapest, Hungary

REFERENCES:
- [Derived] Csukly G, Orban-Szigeti B, Suri K, Zsigmond R, Herman L, Simon V, Kabaji A, Bata B, Harsfalvi P, Vass E, Csibri E, Farkas K, Rethelyi J. Theta-burst rTMS in schizophrenia to ameliorate negative and cognitive symptoms: study protocol for a double-blind, sham-controlled, randomized clinical trial. Trials. 2024 Apr 17;25(1):269. doi: 10.1186/s13063-024-08106-9. PMID 38632647